CLINICAL TRIAL: NCT06774534
Title: The ASSESSMENT of SERPINB3 EXPRESSION, PAR2 and SCCA-PD POLYMORPHISM in PATIENTS with ACUTE RESPIRATORY DISTRESS SYNDROME
Brief Title: SerpinB3 Expression, PAR2 and SCCA-PD Polymorphism in Acute Respiratory Distress Syndrome
Acronym: Serpin-ARDS
Status: Recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Annalisa Boscolo, Professor, University of Padova
Other Study IDs: AOP3543
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Distress Syndrome (RDS); Respiratory Failure
Keywords: ARDS; RESPIRATORY FAILURE; ICU
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CASES: Patients affected by Acute Respiratory Distress Syndrome (ARDS) and needing invasive mechanical ventilation (IMV).
- CONTROLS: Patients admitted to the Intensive Care Unit and requiring IMV not for respiratory reasons.

SUMMARY:
The Acute Respiratory Distress Syndrome (ARDS) is a systemic syndrome characterized by severe respiratory failure, inflammation, loss of aerated tissue and high mortality. Recently, significant efforts have been made to phenotype ARDS patients through a wide range of new biomarkers and imaging indices with the goal of developing personalized treatments based on patient's biophenotypization. Recent literature demonstrates, both in vitro and in vivo but not yet in ARDS patients, that the serine protease inhibitor(SERPIN)-B3 plays a crucial role in the pathological mechanism of pulmonary fibrogenesis, and, similarly, protease-activated receptors(PAR2) is highly involved in this aberrant inflammatory response.

Consequently, studying the expression of SERPINB3 (including SCCA-PD polymorphism) and PAR2, in association with a detailed clinical and biomolecular phenotypization, could allow new insights into the pathophysiological mechanisms of lung injury during ARDS.

DETAILED DESCRIPTION:
SERPINB3 is a strong activator of transforming growth factor-beta (TGF-b), an important pro-fibrogenic cytokine that also promotes epithelial-mesenchymal transition. Its expression can be induced/stimulated by oxidative stress. For example, in patients with idiopathic pulmonary fibrosis, the expression of SERPINB3 is significantly correlated with the presence of severe fibrosis and the expression of TGF-b. Recently, a new polymorphism of SERPINB3 (SCCA-PD) has been identified, featuring a single amino acid substitution in the reactive center loop of the protein, which enhances the functional anti-protease activity of this protein, inducing a more pronounced inflammatory and fibrotic response compared to wild-type SERPINB3, even in cultured monocytic cell lines. However, data is lacking in patients affected by ARDS. Furthermore, the reactive site loop of SERPINB3 has been shown to be essential for activating PAR2, another key element in the pro-fibrogenic cascade. PAR2 belongs to a subfamily of protease-activated G-protein-coupled receptors, consisting of four members, which plays a crucial role not only in activating the coagulation cascade and endothelendothelial inflammation but also in other stress-related clinical responses, such as pulmonary fibrosis. In conclusion, there is currently no data confirming a potential activation of the "SERPINB3-PAR2" pathway in ARDS patient, which is presumably involved in the pathway of severe lung injuries affecting ARDS patients.

More severe hyperinflammatory subphenotypes of ARDS are presumibely correlated with higher expression of SERPINB3, PAR2 and the presence of the SCCA-PD polymorphism. Thus, an early phenotypization of these critically ill patients could:

i) allow the identification and characterization of a subgroup of patients at higher risk of pulmonary fibrosis and death; and, ii) promote the development of new therapeutic strategies, that counteract the fibroproliferative process during ARDS avoiding the activation of "SERPINB3-PAR2" pathway, which could be a new pharmacological target for limiting the aberrant lung injury affecting ARDS patients (see 1-PPA).

Demographic, clinical, and ventilatory data will be collected in accordance with our institutional protocols until hospital discharge. All patients will undergo a high-resolution chest CT scan within 72 hours of ARDS diagnosis using a multidetector CT scan to assess the fibroproliferative changes typical of pulmonary fibrosis. A second high-resolution CT scan will be performed 21 ± 7 days after ARDS diagnosis or at hospital discharge, whichever occurs first, to monitor the evolution of fibroproliferative pulmonary changes.

Blood samples and BAL samples will be collected within 72 hours (and, only if available, at 21 ± 7 days) from ARDS diagnosis, as part of routine clinical practice. Only residual material will be used for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* ARDS DIAGNOSIS
* IMV

Exclusion Criteria:

* Age under 18 years
* Pregnancy status
* Lack of consent to participate in the study
* Contraindications to fiberoptic bronchoscopy and/or BAL (bronchoalveolar lavage)
* Patients with chronic inflammatory skin conditions
* Patients with chronic lung diseases
* Patients with inflammatory respiratory diseases
* Patients with neoplasms such as: squamous cell carcinoma of the cervix, squamous cell carcinoma of the esophagus, lung adenocarcinoma, breast adenocarcinoma, pancreatic adenocarcinoma, hepatocellular carcinoma
* History of active or passive smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients affected by ARDS and requiring IMV
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
SERPINB3 | Within 72 hours from ARDS diagnosis
  Quantifying the expression of SERPINB3, PAR2 (measured in blood, bronchoalveolare lavage (BAL), and extracellular vesicles (EV)) in adult ARDS patients, requiring ventilatory support.
SCCA-PD | Within 72 hours from ARDS diagnosis
  Quantifying the occurrence of SCCA-PD variant in adult ARDS patients, requiring ventilatory support.

SECONDARY OUTCOMES:
FIBROSIS and SERPINB3, PAR2, SCCA-PD variant | At 21 days from ARDS diagnosis
  Investigating potential correlations between the Ichikado score (calculated on the CTscan performed after 21±7 days from ARDS diagnosis) and the expression of SERPINB3, PAR2 and the SCCA-PD variant.
60-DAY MORTALITY PREDICITVE MODELS | At 60-day after ARDS diagnosis
  Subsequently, identifying new models able to predict 60-day mortality according to anthropometric, clinical, respiratory parameters and laboratory data of lung damage (i.e., SERPINB3, PAR2, inflammatory cytokines (including TNF-a, TGF-ß ect) and cytofluorimetric measurements).

OTHER OUTCOMES:
Only if available | At 21 days after ARDS diagnosis
  Quantifying the expression of SERPINB3, PAR2 (measured in blood, bronchoalveolare lavage (BAL), and extracellular vesicles (EV)) in adult ARDS patients, requiring ventilatory support.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Padova, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Undecided